CLINICAL TRIAL: NCT03584919
Title: Comparison of Doxycycline and Cefuroxime Axetil in Patients With Erythema Migrans
Brief Title: Comparison of Doxycycline and Cefuroxime Axetil in Erythema Migrans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Daša Stupica, Principal Investigator, University Medical Centre Ljubljana
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Doxy-Zinnat
Record Dates: First submitted 2018-06-19; First posted 2018-07-12 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-06

CONDITIONS: Erythema Chronicum Migrans
MeSH Terms: conditions — Erythema Chronicum Migrans | interventions — Doxycycline; cefuroxime axetil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EM doxycycline (Active Comparator): patients with EM who received doxycycline
  Interventions: Drug: doxycycline
- EM cefuroxime axetil (Active Comparator): patients with EM who received cefuroxime axetil
  Interventions: Drug: Cefuroxime Axetil 500Mg Tab
- controls (Placebo Comparator): control subjects without history of Lyme disease
  Interventions: Other: control subjects

INTERVENTIONS:
Drug: doxycycline — patients received oral doxycycline 100 milgrams bid for 15 days
  Arms: EM doxycycline
Drug: Cefuroxime Axetil 500Mg Tab — patients received cefuroxime axetil 500 milgrams bid for 15 days
  Arms: EM cefuroxime axetil
Other: control subjects — no intervention
  Arms: controls

SUMMARY:
A European, prospective clinical trial in which doxycycline and cefuroxime axetil were compared in the treatment of adult patients with erythema migrans included a control group to address this question. Evaluations of patients were conducted at baseline, 14 days and 2, 6, and 12 months after enrollment. Control subjects were evaluated at baseline and at 6 and 12 months. Subjective complaints that newly developed or intensified since the onset of erythema migrans or since the date of enrollment for controls were referred to as "new or increased symptoms"(NOIS).

ELIGIBILITY:
Inclusion Criteria:

* typical solitary erythema migrans as defined by the United States Centers for Disease Control and Prevention. In addition, patients with skin lesion <5 cm in diameter were also included if they recalled a recent tick bite at the site of the skin lesion, had a symptom-free interval between the bite and the onset of the lesion, and reported an expanding skin lesion prior to diagnosis.

Exclusion Criteria:

* Lyme disease previously
* pregnancy or lactation
* immunocompromised
* serious adverse reaction to a beta-lactam or tetracycline drug in the past
* received an antibiotic with known anti-borrelial activity within 10 days
* multiple erythema migrans lesions
* presence of an extracutaneous manifestation of Lyme disease

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 509
Dates: Start 2006-06-01 (Actual); Primary Completion 2007-09-30 (Actual); Study Completion 2007-09-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Objective Manifestations and Subjective New or Increased Symptoms (NOIS) in Patients Treated for Erythema Migrans With Doxycycline or Cefuroxime Axetil for 15 Days | One year follow-up (follow-up time points at 14 days, 2 months, 6 months, and 12 months after enrolment)
  At each visit patients were examined and asked about the presence of any symptoms that newly developed or had worsened since erythema migrans. If such symptoms had no other medical explanation they were regarded as new or increased symptoms (NOIS). Complete response was defined as absence of any manifestations of Lyme borreliosis, with return to pre-Lyme borreliosis health status. Partial response was defined as presence of NOIS. Failure was defined as presence of objective manifestations of Lyme borreliosis or persistence of Borrelia burgdorferi sensu lato in skin at the site of the previous erythema migrans.

SECONDARY OUTCOMES:
Number of Patients (at 12 Months After Treatment With Doxycycline or Cefuroxime Axetil for 15 Days for Erythema Migrans) and Number of Control Subjects (Without a History of Lyme Borreliosis) With Nonspecific Symptoms. | 12 months after treatment
  12 months after treatment patients and controls were asked to complete a written questionnaire asking whether they had had any of 8 nonspecific symptoms (fatigue, arthralgias, headache, myalgias, paresthesias, concentration difficulties, or irritability) within the preceding week. For both patients and controls, the severity of each individual symptom was graded by the subject on a 10-cm visual analog scale (10 = most severe).

REFERENCES:
- [Derived] Veluscek M, Bajrovic FF, Strle F, Stupica D. Doxycycline-induced photosensitivity in patients treated for erythema migrans. BMC Infect Dis. 2018 Aug 3;18(1):365. doi: 10.1186/s12879-018-3270-y. PMID 30075748